CLINICAL TRIAL: NCT00334061
Title: Evaluation of the Penumbra™ Stroke System in the Revascularization of Patients With Acute Ischemic Stroke Secondary to Intracranial Large Vessel Occlusive Disease
Brief Title: Study to Assess the Safety and Effectiveness of the Penumbra System
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Penumbra Inc. (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLP 0676
Record Dates: First submitted 2006-06-02; First posted 2006-06-06 (Estimated); Results first posted 2009-01-12 (Estimated); Last update posted 2019-09-18 (Actual); Status verified 2019-09

CONDITIONS: Stroke
Keywords: Penumbra; Ischemic; Stroke; Intervention; Neurovascular; Thrombus; Embolectomy; Ischemic stroke
MeSH Terms: conditions — Stroke; Ischemia; Thrombosis; Ischemic Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: Penumbra System

SUMMARY:
This clinical evaluation is a prospective, single-arm, multi-center trial.

The purpose of this clinical evaluation is to assess the safety and effectiveness of the Penumbra System in the revascularization of patients presenting with acute ischemic stroke secondary to intracranial, large vessel, occlusive disease.

DETAILED DESCRIPTION:
Purpose:

The purpose of this clinical evaluation is to assess the safety and effectiveness of the Penumbra System in the revascularization of patients presenting with acute ischemic stroke secondary to intracranial, large vessel, occlusive disease. Up to 125 evaluable patients will be enrolled in the study.

ELIGIBILITY:
Inclusion Criteria:

* Clinical signs consistent with acute ischemic stroke
* 18 to 79 years of age
* Neurological deficit resulting in an NIH Stroke Scale (NIHSS) score > 8
* TIMI 0 or TIMI I flow in vessels accessible to the Penumbra System
* Signed informed consent
* Present within 8 hours of stroke symptom onset; ineligible or refractory to intravenous tissue plasminogen activator (t-PA) therapy if presenting within 3 hours of symptom onset.

Exclusion Criteria:

* Evidence of rapidly improving neurological signs of stroke at time of enrollment
* NIHSS > 30 or coma
* Females who are pregnant
* Vessel tortuosity too difficult to allow endovascular access
* Known hemorrhagic diathesis, coagulation deficiency, or on oral anticoagulant therapy with an International Normalized Ratio (INR) > 3.0
* Partial thromboplastin time (PTT) greater than 2 times the lab normal
* Admission platelets < 30,000
* Pre-existing neurological or psychiatric disease that could confound the study results
* Known severe allergy to contrast media
* Uncontrolled hypertension
* Computed tomography (CT) evidence of significant mass effect with a midline shift
* CT reveals evidence of large hypodensity region > 1/3 of the middle cerebral artery territory
* CT reveals evidence of intracranial hemorrhage
* CT reveals significant mass effect with midline shift
* Angiographic evidence of an arterial stenosis proximal to the occlusion that could prevent thrombus removal
* Angiographic evidence of preexisting arterial injury
* Life expectancy of less than 90 days
* Participation in another clinical investigation that could confound the evaluation of the study device.

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125 (Actual)
Dates: Start 2006-06; Primary Completion 2007-06 (Actual); Study Completion 2007-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Saint Luke's Hospital, Kansas City, Missouri, United States

REFERENCES:
- See also: Related Info — http://www.penumbrainc.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: From June 19, 2006 to June 5, 2007 a total of 856 patients were screened of which 125 patients were enrolled at 24 centers in Europe and the United States.
Period: Overall Study
Arm/Group | Penumbra System
Started | 125 (June 2006)
Completed | 125 (November 2007)
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Penumbra System
Number analyzed (Participants) | 125
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1
  Between 18 and 65 years | 53
  >=65 years | 71
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.5 (13.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 61
  Male | 64
Region of Enrollment [Number; unit: participants]
  United States | 76
  Europe | 49

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Revascularization of the Occluded Target Vessel
Description: Revascularization is defined by a Thrombolysis in Myocardial Infarction (TIMI) score of 2 or 3 following use of the Penumbra System.
  TIMI scores are used to describe blood flow at the treated vessel with 0 designating no flow and 3 for normal flow.
Time Frame: 3-Month Post-Procedure
Population: Intention to Treat
Measure: Number; unit: Percentage of Participants
Arm/Group | Penumbra System
Number analyzed (Participants) | 125
Percentage of Participants | 81.2

2. Primary Outcome: Percentage of Participants With Device-related and Procedure-related Serious Adverse Events
Time Frame: 3-Month Post-Procedure
Population: All adverse events were summarized by showing the number and percent of patients who reported the event. Events were also reported by relationship to the procedure or device. Causality of adverse events was adjudicated by a Clinical Events Committee. The denominator for the analyses was all enrolled patients.
Measure: Number; unit: Percentage of Participants
Arm/Group | Penumbra System
Number analyzed (Participants) | 125
Percentage of Participants | 2.4

3. Secondary Outcome: Percentage of Participants With Either a 4-point Improvement on the National Institutes of Health Stroke Scale (NIHSS) at Discharge or a Modified Rankin Scale (mRS) Score of ≤ 2 at 30 Days After Treatment
Description: NIHSS is a 42 point scale to describe the neurological status of the patients:
  0=no stroke; 1-15=minor to moderate stroke; 15-20=moderate/severe stroke; 21-42=severe stroke. The mRS is a scale to determine the activities of daily living of the patient with a score of 0 designating normal activities to a score of 6 designating death.
Time Frame: Discharge or 30-Days Post-Procedure
Measure: Number; unit: Percentage of Participants
Arm/Group | Penumbra System
Number analyzed (Participants) | 125
Percentage of Participants | 41.6

4. Secondary Outcome: Percentage of Participants With a Modified Rankin Scale (mRS) Score of ≤ 2 at 90 Days Post Treatment
Description: The mRS is a scale to determine the activities of daily living of the patient with a score of 0 designating normal activities to a score of 6 designating death.
Time Frame: 90-Day
Measure: Number; unit: Percentage of Participants
Arm/Group | Penumbra System
Number analyzed (Participants) | 125
Percentage of Participants | 25

5. Secondary Outcome: Percentage of Participants With All Cause Mortality
Time Frame: 90-Days Post-Treatment
Measure: Number; unit: Percentage of Participants
Arm/Group | Penumbra System
Number analyzed (Participants) | 125
Percentage of Participants | 32.8

6. Secondary Outcome: Percentage of Participants With Symptomatic Hemorrhage
Description: All treated patients were scanned by computed tomography (CT) at 24-hours post-procedure to detect the presence of intracranial hemorrhage.
Time Frame: 24-Hour Post-Procedure
Measure: Number; unit: Percentage of Participants
Arm/Group | Penumbra System
Number analyzed (Participants) | 125
Percentage of Participants | 11.2

ADVERSE EVENTS:
Arm/Group | Penumbra System
Serious Adverse Events (participants affected / at risk) | 65/125
Other Adverse Events (participants affected / at risk) | 125/125
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Penumbra System (N=125)
Cerebral Edema (Nervous system disorders) | 14
Intracerebral Hemorrhage (Nervous system disorders) | 10
Respiratory Dysfunction/Failure (Respiratory, thoracic and mediastinal disorders) | 10
Worsening Symptoms of Qualifying Stroke (Nervous system disorders) | 9
Infection (General disorders) | 7
Other Pulmonary Complications (Respiratory, thoracic and mediastinal disorders) | 7
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 5
Cardiac Arrhythmia (Cardiac disorders) | 4
Access Site Complication (Skin and subcutaneous tissue disorders) | 3
Myocardial Infarction (Cardiac disorders) | 3
Peripheral Vascular Complication (Vascular disorders) | 3
Renal Dysfunction/Failure (Renal and urinary disorders) | 3
Stroke in New Territory (Nervous system disorders) | 3
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Penumbra System (N=125)
Infection (Infections and infestations) | 31
Pneumonia (Infections and infestations) | 23
Electrolyte Imbalance (Metabolism and nutrition disorders) | 22
Pain (General disorders) | 21
Fever (General disorders) | 14
Anemia (Blood and lymphatic system disorders) | 13
Cardiac Arrhythmia (Cardiac disorders) | 13
Cerebral Edema (Injury, poisoning and procedural complications) | 12
Other Pulmonary Complications (Respiratory, thoracic and mediastinal disorders) | 12
Hyperglycemia (Hepatobiliary disorders) | 10
Hypotension (Vascular disorders) | 9
Nausea (Gastrointestinal disorders) | 9
Headache (Nervous system disorders) | 8
Peripheral Vascular Complication (Vascular disorders) | 8
Constipation (Gastrointestinal disorders) | 7
Renal Dysfunction/Failure (Renal and urinary disorders) | 7
Coagulopathy (Blood and lymphatic system disorders) | 5
Depression (Psychiatric disorders) | 5
Hepato-Biliary Dysfunction (Hepatobiliary disorders) | 5
Peripheral Edema (Metabolism and nutrition disorders) | 5
Worsening Symptoms of Qualifying Stroke (Nervous system disorders) | 5
Dysphasia-Aspiration (Psychiatric disorders) | 4
Hypertension (Vascular disorders) | 4
Peripheral Hemorrhage (Vascular disorders) | 4
Anxiety (Psychiatric disorders) | 3
Cardiac Complications (Cardiac disorders) | 3
Confusion (Psychiatric disorders) | 3
Diarrhea (Gastrointestinal disorders) | 2
Embolization of Previously Uninvolved Vessel (Vascular disorders) | 2
GERD (Gastrointestinal disorders) | 2
Seizure (Nervous system disorders) | 2
Ulcer (General disorders) | 2
Other (General disorders) | 16

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less